CLINICAL TRIAL: NCT02921893
Title: Ixazomib, Lenalidomide, and Dexamethasone for Patients With POEMS Syndrome
Brief Title: Ixazomib Citrate, Lenalidomide, and Dexamethasone in Treating Patients With POEMS Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1682; NCI-2016-01426 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1682 (Other: Mayo Clinic in Rochester); 16-002976 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2016-09-26; First posted 2016-10-03 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Plasmacytoma; POEMS Syndrome
MeSH Terms: conditions — Plasmacytoma; POEMS Syndrome | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ixazomib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (ixazomib citrate, lenalidomide, dexamethasone, ASCT) (Experimental): Patients receive ixazomib citrate PO on days 1, 8, and 15, lenalidomide PO QD on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo standard of care ASCT after completing 3 cycles of treatment.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib Citrate; Drug: Lenalidomide; Other: Questionnaire Administration
- Group II (ixazomib citrate, lenalidomide, dexamethasone) (Experimental): Patients receive ixazomib citrate PO, lenalidomide PO QD, and dexamethasone PO as in Group I. Treatment repeats every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib Citrate; Drug: Lenalidomide; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well ixazomib citrate, lenalidomide, and dexamethasone work in treating patients with polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome. Ixazomib citrate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Anti-inflammatory drugs, such as dexamethasone lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Giving ixazomib citrate, lenalidomide, and dexamethasone may work better in treating patients with POEMS syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Normalization of VEGF after 3 cycles of therapy.

SECONDARY OBJECTIVES:

I. Toxicity and safety of the combination of ixazomib citrate (ixazomib), lenalidomide, and dexamethasone.

II. Hematologic response after 3 cycles of therapy. III. Hematologic response rates and/or VEGF response at 12 months. IV. Overall survival.

EXPLORATORY OBJECTIVES:

I. Improvement of peripheral neuropathy (Overall Neuropathy Limitations Scale [ONLS], Modified Neurological Impairment Score for POEMS [mNIS+7POEMS], and performance score), ascites/effusions, diffusing capacity of the lungs for carbon monoxide (DLCO) after 3 cycles of therapy.

II. Improvement of peripheral neuropathy (ONLS, mNIS+7POEMS, and performance score), ascites/effusions, DLCO, and positron emission tomography (PET)-scan (if abnormal at baseline) at 12 months (both groups) and at 24 and 36 months (group 2 only).

III. Time to VEGF response, hematologic response, and clinical response. IV. Time to VEGF progression, hematologic progression, and clinical progression.

V. Doses delivered will be tabulated to establish tolerance of study drugs.

CORRELATIVE RESEARCH OBJECTIVES:

I. To describe changes in bone biomarkers with treatment of ixazomib, lenalidomide, and dexamethasone.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I: Patients receive ixazomib citrate orally (PO) on days 1, 8, and 15, lenalidomide PO once daily (QD) on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo standard of care autologous stem cell transplant (ASCT) after completing 3 cycles of treatment.

GROUP II: Patients receive ixazomib citrate PO, lenalidomide PO QD, and dexamethasone PO as in Group I. Treatment repeats every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months until disease progression and then every 6 months for up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* POEMS syndrome requiring therapy, previously treated or untreated
* Plasma vascular endothelial growth factor (VEGF) > 2 x upper limit of normal (ULN)
* Presence of a plasma cell clone (any of the following):

  * Monoclonal protein in the serum or urine
  * Measurable light chains by free light chain assay
  * Measurable plasmacytoma
  * Monoclonal plasma cells in bone marrow
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, 2, or 3
* Absolute neutrophil count (ANC) >= 1000/uL obtained =< 14 days prior to registration
* Platelet count (PLT) >= 75,000/uL obtained =< 14 days prior to registration
* Total bilirubin =< 2.0 mg/dL unless due to known Gilbert's disease obtained =< 14 days prior to registration

  * NOTE: If total bilirubin is > 2 mg/dL, a direct bilirubin should be performed and must be < 1.5 mg/dL for Gilbert's to be diagnosed
* Alanine aminotransferase (ALT/serum glutamic pyruvic transaminase [SGPT]) and aspartate aminotransferase (AST, serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x upper limit of normal (ULN) obtained =< 14 days prior to registration
* Creatinine clearance >= 30 mL/min/1.73 m^2 (as determined by Cockcroft-Gault equation) obtained =< 14 days prior to registration
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only

  * NOTE: Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid Risk Evaluation and Mitigation Strategy (REMS) program
* Birth control

  * Female patients of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication

    * NOTE: Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
  * Male patients must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

    * NOTE: Abstinence is acceptable (for either males or females) if this is the established and preferred method of contraception for the subject
* Willing to adhere to the guidelines of the Revlimid REMS (formerly known as RevAssist) program

  * NOTE: The counseling must be documented
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

  * Note: During the active monitoring phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* No contraindication to be on a minimum of 81 mg aspirin a day (or other anticoagulant therapy as prescribed) for thromboembolism prophylaxis
* Willing to provide mandatory blood and bone marrow samples for research purposes
* Ability to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

* Recent prior chemotherapy:

  * Newly diagnosed patients (regardless of group); any prior chemotherapy for POEMS with the following exceptions:

    * Prior immunomodulators like azathioprine, cyclosporin, and/or corticosteroids are not exclusionary therapies if used for prior diagnosis of chronic inflammatory demyelinating polyneuropathy
    * Prior chemotherapy directed at a "myeloproliferative neoplasm" like hydroxyurea is not exclusionary
  * Previously treated patients (group 2)

    * Alkylators (e.g. melphalan, cyclophosphamide) =< 28 days prior to registration
    * Anthracyclines =< 28 days prior to registration
    * High dose corticosteroids, immune modulatory drugs (thalidomide or lenalidomide), or proteosome inhibitors (e.g. ixazomib or bortezomib) =< 28 days prior to registration
* Requirement for concomitant high dose corticosteroids

  * EXCEPTION: Patients may be on chronic steroids (maximum dose 20 mg/day prednisone equivalent) if they are being given for adrenal insufficiency, rheumatoid arthritis, etc
* Receiving any other investigational agent, which would be considered as a treatment for the primary neoplasm
* Participation in other clinical trials, including those with other investigational agents not included in this trial, =< 30 days prior to registration and throughout the duration of this trial
* Prior refractoriness to proteasome inhibitor or immunomodulatory drugs (IMiD)
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other active malignancy =< 3 years prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer, ductal carcinoma in-situ, or carcinoma-in-situ of the cervix
  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens, e.g. uncontrolled infection (infection requiring systemic antibiotic therapy or other serious infection =< 14 days prior to registration); or uncompensated heart or lung disease
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy
* Systemic treatment with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort =< 14 days prior to registration
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Radiotherapy =< 14 days prior to registration
* Major surgery =< 14 days prior to registration
* Failure to fully recover (i.e. =< grade 1 adverse event [AE]) from the reversible effects of prior chemotherapy
* Known allergy to any of the study medications, their analogs, or excipients in the various formulations of any agent
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of the study drugs including difficulty swallowing
* Ongoing or active systemic infection or active hepatitis B or C virus infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Rate of normalization of VEGF defined as VEGF value decreasing to below upper limit of normal (86 pg/mL) | Up to 3 months
  In each group, the rate of normalization of VEGF by 3 months (post-3 cycles) will be examined along with the prognostic factors for patients accrued to this study. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent binomial confidence intervals for the true success proportion will be calculated.

SECONDARY OUTCOMES:
Hematologic response rate | Up to 3 months
  Hematologic response rate after 3 cycles of therapy (or 3 months after registration) will be estimated by the number of hematologic responses (partial response, very good partial response, or complete response) observed within 3 months of registration divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true hematologic response rate after 3 cycles of therapy (or 3 months after registration) will be calculated.
Hematologic response rate | Up to 12 months
  Hematologic response rate after 13 cycles of therapy (or 12 months) will be evaluated. Exact binomial 95% confidence intervals for the true rates at 12 months will be calculated.
Normalization of VEGF | Up to 12 months
  Normalization of VEGF after 13 cycles of therapy (or 12 months after registration) will be evaluated. Exact binomial 95% confidence intervals for the true rates at 12 months will be calculated.
Survival time | Time from registration to death due to any cause, assessed up to 3 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Incidence of adverse events evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 3 years
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

OTHER OUTCOMES:
Change in peripheral neuropathy evaluated by Modified Neurological Impairment Score +7 polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes | Baseline up to 36 months
  Improvement of peripheral neuropathy (Modified Neurological Impairment Score +7 polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) will be defined as decrease of >= 2 points. Other neurologic tests including Overall Neuropathy Limitations Scale, polyneuropathy disability score, and EQ-5D-5L health questionnaire will be analyzed descriptively.
Change in positron emission tomography-scan | 3 months up to 36 months
  Improvements will be assessed by evaluating changes from baseline and will be described descriptively.
Change in presence or absence of ascites/effusions/edema | 3 months up to 36 months
  Improvements will be assessed by evaluating changes from baseline and will be described descriptively.
Change in right ventricular systolic pressure evaluated by echocardiogram | 3 months up to 36 months
  Improvements will be assessed by evaluating changes from baseline and will be described descriptively.
Change in diffusion capacity of the lung for carbon monoxide | 3 months up to 36 months
  Improvements will be assessed by evaluating changes from baseline and will be described descriptively.
Change in presence or absence of papilledema | 3 months up to 36 months
  Improvements will be assessed by evaluating changes from baseline and will be described descriptively.
Time to VEGF response | Time from registration to the time of response, assessed up to 3 years
  Median and range will be calculated for time to response in responding patients.
Time to hematologic response | Time from registration to the time of response, assessed up to 3 years
  Median and range will be calculated for time to response in responding patients.
Time to clinical response | Time from registration to the time of response, assessed up to 3 years
  Median and range will be calculated for time to response in responding patients.
Time to VEGF progression | Time from registration to the time of progression, assessed up to 3 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time to hematologic progression | Time from registration to the time of progression, assessed up to 3 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time to clinical progression | Time from registration to the time of progression, assessed up to 3 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Drug tolerance | Up to 3 years
  Doses delivered will be tabulated to establish tolerance of drugs. Reasons for dose adjustments will be evaluated. Dose levels by cycle and total dose will be evaluated and summarized using descriptive statistics (median, range).
Change in bone biomarkers procollagen type I N propeptide and collagen type 1 C-telopeptide | Baseline to 36 months
  Will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials